CLINICAL TRIAL: NCT03993938
Title: Pleth Variability Index (PVI) as a Measure of Volume Status During Transcatheter Mitral Valve Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Ashwin Vaidyanathan, MD, Principal Investigator, Resident, Department of Anesthesiology, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1
Record Dates: First submitted 2019-02-17; First posted 2019-06-21 (Actual); Results first posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-05

CONDITIONS: Mitral Regurgitation
Keywords: transcatheter mitral valve repair; pleth variability index; Mitraclip
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Patients for TMVR (Experimental): Patients with severe mitral regurgitation scheduled for TMVR procedure at Henry Ford Hospital - main campus.
  Interventions: Device: PVI measurement

INTERVENTIONS:
Device: PVI measurement — Masimo Radical-7® probe to be attached to patient's finger along with standard ASA monitors at the start of procedure. After placement of arterial line, stroke volume variation (SVV) and pulse pressure variation (PPV) to be recorded along with pleth variability index (PVI) every 5 minutes. Intraprocedure left atrial pressure (LAP) (v-wave and mean) to be recorded prior to and after MitraClip deployment. Data to be analyzed - age, sex, BMI; Preprocedure ejection fraction (EF), pulmonary artery pressure (PAP), rhythm, mitral regurgitation severity; heart rate, systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial pressure (MAP) every 5 minutes; SVV, PPV, PVI every 5 minutes; LAP prior to mitraclip deployment; LAP after mitraclip deployment

SUMMARY:
Transcatheter mitral valve repair in the form of MitraClip® is a safe and effective alternative to surgical mitral valve repair/replacement in patients with high operative morbidity and mortality risk. Successful MitraClip application depends on intraprocedural quantification of mitral regurgitation and left atrial pressure (LAP) monitoring. The pleth variability index (PVI) is a noninvasive, dynamic index based on analysis of the respiratory variations in the plethysmographic waveform recorded transcutaneously by the pulse oximeter. Studies demonstrate that PVI is accurate in predicting fluid responsiveness in mechanically ventilated adult patients. In this study, we wish to measure PVI during TMVR and correlate with invasive indices such as left atrial pressure (LAP) and stroke volume variation. Our study hopes to provide a real-time non-invasive alternative to invasive indices to better guide fluid management and improve hemodynamics.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with mitral regurgitation undergoing transcatheter mitral valve repair(TMVR) with Mitra-Clip(R) at Henry Ford Hospital - Main Campus.

Exclusion Criteria:

* MitraClip(R) procedure unsuccessful (defined as no clip deployment and/or procedural interruption due to complication), concomitant aortic regurgitation or stenosis of moderate or greater degree existed, patients with grade II or above diastolic dysfunction on echocardiography, previous mitral valve intervention (either surgical or percutaneous), patients requiring continuous vasopressor infusions during the procedure, or patients in whom PVI monitoring was not performed due to technical issues, patients with atrial fibrillation, or preprocedure moderate or greater mitral stenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vaidyanathan A, Guruswamy J, Saluja A, Eng M, Szymanski T. Use of Pleth Variability Index as a Non-invasive, Dynamic Indicator of Left Atrial Pressure Change During MitraClip: Transcatheter Mitral Valve Repair. Semin Cardiothorac Vasc Anesth. 2024 Sep;28(3):147-151. doi: 10.1177/10892532241260535. Epub 2024 Jun 12. PMID 38864441

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients for TMVR
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients for TMVR
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 25
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 80 [77 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 23
  More than one race | 0
  Unknown or Not Reported | 1
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 25.4 [23.2 to 29.2]
Ejection fraction [Median (Inter-Quartile Range); unit: %] | 47.5 [31.2 to 57.2]
Mean pulmonary artery (PA) pressure [Median (Inter-Quartile Range); unit: mm Hg] | 43 [33 to 51]

OUTCOME MEASURES:

1. Primary Outcome: Delta PVI to Delta LAP Correlation During MitraClip Placement
Description: Delta pleth variability index (PVI) and delta left atrial pressure (LAP) are calculated by subtracting the values of LAP (as obtained intraprocedurally) and corresponding PVI value (as recorded by the Masimo Radical-7 probe) from the LAP and PVI value respectively after MitraClip placement. The delta PVI and delta LAP for the sample patient population are correlated to obtain the Pearson correlation coefficient and p-value
Time Frame: Intraprocedure
Measure: Median (Inter-Quartile Range); unit: percentage of baseline (pre-MitraClip)
Arm/Group | Patients for TMVR
Number analyzed (Participants) | 30
percentage of baseline (pre-MitraClip)
  Delta PVI (percentage change) | 4.30 [-15.06 to 40.91]
  Delta LAP (percentage change) | -26.14 [-42.36 to -11.46]
Statistical Analysis 1: Comparison: Patients for TMVR; Test type: Other — Delta PVI percentage change and Delta LAP (v-wave) percentage change were correlated using Spearman's rank correlation - two-tailed; p = 0.066, Spearman's rank correlation; Spearman's rank correlation = 0.34

ADVERSE EVENTS:
Time Frame: 1 year 4 months
Arm/Group | Patients for TMVR
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-30): https://cdn.clinicaltrials.gov/large-docs/38/NCT03993938/Prot_SAP_000.pdf